CLINICAL TRIAL: NCT04034550
Title: Cohort of Hospitalized Patients Suspected of Leptospirosis
Acronym: COLEPT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: C17-47
Record Dates: First submitted 2019-07-25; First posted 2019-07-26 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Leptospirosis
Keywords: leptospirosis; hospitalization
MeSH Terms: conditions — Leptospirosis | interventions — Blood Specimen Collection; Blood Banking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hospitalized patients diagnosed with leptospirosis (Experimental): hospitalized patients diagnosed with leptospirosis: 12 months of follow up with biological samples and data collection
  Interventions: Other: Blood and urine sampling and blood banking

INTERVENTIONS:
Other: Blood and urine sampling and blood banking — In routine management, blood and urine will be sampled for each patients and specific analyses carried out. Only blood samples will be banked.

SUMMARY:
COLEPT is a prospective interventional study that intends to better inform about leptospirosis, a neglected zoonotic infectious disease. During prospective follow-up of hospitalized acute leptospirosis cases, the participants will be assessed during 1 year for epidemiological, clinical, bacteriological and immunological data. Main intervention consists in blood sampling and biological bank constitution.

ELIGIBILITY:
Inclusion Criteria:

* clinico-biological manifestations compatible with acute leptospirosis OR proven leptospirosis with serological testing or PCR
* onset of symptoms within 21 days
* participant benefits of health insurance

Exclusion Criteria:

* participant's refusal, or refusal from his relatives in case of major incapacity of the eligible participant precluding expression of his will (coma, stay in intensive care unit))

Min Age: 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-01-06 (Actual); Primary Completion 2027-01-06 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
disease severity | 0 to 21 days after onset of symptoms
  Rate of death or severe organ insuffisiency

CONTACTS AND LOCATIONS:
Overall Officials: Loïc RAFFRAY, MD, PhD, Principal Investigator — CHU Reunion, INSERM, CNRS, IRD UMR PIMIT
Locations (4):
- France (4):
  - Groupe Hospitalier Est Réunion (GHER), Saint-Benoît, Reunion
  - CHU de La Réunion site Nord, Saint-Denis, Reunion
  - Centre Hospitalier Ouest Réunion (CHOR), Saint-Paul, Reunion
  - CHU de La Réunion site Sud (GHSR), Saint-Pierre, Reunion